CLINICAL TRIAL: NCT03219385
Title: Directed Ablation of Uterine Fibroids Using a Noninvasive Approach (DIANA)
Brief Title: Directed Ablation of Uterine Fibroids Using a Noninvasive Approach
Acronym: DIANA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mirabilis Medica, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMI 2001
Record Dates: First submitted 2017-07-13; First posted 2017-07-17 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Uterine Leiomyoma
Keywords: uterine leiomyoma; uterine fibroid; uterine myoma; abnormal menstrual bleeding; heavy menstrual bleeding; menorrhagia; high-intensity focused ultrasound; ultrasound imaging
MeSH Terms: conditions — Myofibroma; Leiomyoma; Menorrhagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment with the Mirabilis System (Experimental)
  Interventions: Device: Mirabilis System

INTERVENTIONS:
Device: Mirabilis System — The intervention is a transabdominal treatment performed with the Mirabilis System, during which high-intensity focused ultrasound (HIFU) is applied noninvasively through the skin using an applicator placed against the abdomen. One or more appropriately selected uterine fibroids will be treated with HIFU using integrated ultrasound imaging to guide the treatment. HIFU causes localized heating and mechanical effects to develop in the targeted fibroid(s) that result in therapeutic destruction of the fibroid tissue, leading to improvement in related symptoms.

SUMMARY:
The purpose of this clinical study is to assess the safety and effectiveness of the Mirabilis System for treating uterine fibroids in women who are seeking relief from fibroid-related abnormal uterine bleeding but want to avoid hysterectomies or other surgical procedures. The Mirabilis System is an investigational device that delivers high-intensity focused ultrasound (HIFU) to the uterus using integrated ultrasound imaging guidance to offer noninvasive treatment for uterine fibroids. With the Mirabilis System, HIFU is applied noninvasively through the skin using an applicator that is placed against the abdomen. No incisions or surgical procedures are required. During this study, eligible patients will have one or more fibroids treated with the Mirabilis System and will then remain in the study for a total of 36 months after treatment to monitor the occurrence of adverse events. Primary endpoints will be assessed at 12 months after treatment, while secondary endpoints will be assessed at variable times ranging from immediately after treatment up to 36 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients between the ages of 18 to 50 years of age.
2. Patients must have 1-3 treatable fibroids with at least one distorting the endometrial cavity.
3. Patients must have at least 1 treatable fibroid or cluster of fibroids that measures between 2 cm to 7 cm in diameter with diagnostic ultrasound.
4. Patients must have primary complaint of prolonged and/or heavy menstrual bleeding.
5. Patients must be in generally good health and seeking relief of fibroid related symptoms.
6. Patients must have a normal Pap smear within 36 months of enrollment, including an endometrial biopsy, if clinically indicated.
7. Patients must be willing to adhere to the study schedule.
8. Patients must have a baseline Menstrual Pictogram (MP) score between 150 mL and 500 mL.
9. Patients must agree to abstain from having other treatments or therapies for fibroids, including procedures (i.e. uterine artery embolization, hysterectomy, radiofrequency ablation of fibroids, etc.) or medications (i.e. hormone therapy for treatment of fibroids; prescription or over the counter medications, including standard, homeopathic, or naturopathic medications, for the treatment of fibroids; dietary supplements taken for the treatment of fibroids, etc.). Exceptions include the use of analgesics or other pain control medications.
10. Patients must have regular cyclical menstrual periods.
11. Patients must be willing to maintain use of their current form of birth control during screening and for 12 months after treatment.
12. Patients must be willing and able to consent to participate in the study.

Exclusion Criteria:

1. Patients who are pregnant, suspected to be pregnant, or wish to become pregnant.
2. Patients unable or unwilling to use only the sanitary products provided by Sponsor during their participation in the study.
3. Patients with fibroids that are deeper than the maximal treatment depth of the Mirabilis System.
4. Patients with fibroids that have certain MRI characteristics including:

   1. A hyper-intense appearance on T2-weighted MRI where the fibroid tissue appears brighter than surrounding myometrium
   2. Features consistent with high perfusion, low perfusion, non-perfusion, infarct, or ischemia on gadolinium-enhanced MRI
   3. Features consistent with extensive degeneration
   4. Fibroids are not quantifiable on MRI
   5. Any endometrial polyp 1 cm or larger
   6. Type 0 fibroids (pedunculated intracavitary)
5. Patients with known endometrial hyperplasia.
6. Patients planning or seeking additional therapies for the treatment of fibroids and/or abnormal uterine bleeding.
7. Patients with other pelvic masses of unknown etiology.
8. Patients who are postmenopausal.
9. Patients with an active diagnosis of cancer of any type.
10. Patients on hormone therapy such as Depo-Provera, Lupron, etc.
11. Patients who within 6 months prior to enrollment had procedures or surgery for the fibroid(s) to be treated as part of this clinical study.
12. Patients with known or suspected bleeding disorders.
13. Patients currently taking anticoagulant therapy.
14. Patients with anemia (hematocrit < 30).
15. Patients with known or suspected endometriosis, adenomyosis, endometrial hyperplasia, and/or active pelvic infection.
16. Patients with visible or suspected scars that are likely to be in the potential HIFU beam path.
17. Patients with an IUD or other implants that cannot be removed from the potential HIFU beam path prior to treatment.
18. Patients who have sensory loss or dysesthesia in the area to be treated.
19. Patients with a history of abdominoplasty or liposuction in the potential HIFU beam path.
20. Patients who currently use illicit drug(s) or abuse alcohol (defined as regular consumption of ≥ 4 alcoholic drinks per day).
21. Patients participating in other clinical studies, except observational or registry studies.
22. Patients unable to tolerate gadolinium enhanced MRI procedures.
23. Patients with significant systemic disease.
24. Patients with known or suspected adhesions in the HIFU beam path. This includes patients who have had abdominoplasty, multiple abdominal surgeries, documented abdominal or pelvic adhesions observed during any prior laparotomy or laparoscopy, surgical mesh placement in the lower abdomen, abdominal abscess such as ruptured appendicitis and tubo-ovarian abscess, or multiple liposuction procedures of the lower abdomen.
25. Patients who cannot or are unlikely to adhere to the study schedule.
26. Patients with a significant psychiatric condition.
27. Patients who lack the capacity to self-consent.
28. Patients with chronic steroid use.
29. Patients on immunosuppressive therapy.
30. Inadequate ultrasound image quality during pre-treatment planning or treatment delivery.
31. The uterus size does not allow the Safety Margin to fit entirely within the uterus while the Target Volume is positioned on the fibroid to be treated.
32. Bowel, bladder, bone, or other sensitive tissue cannot be removed from or avoided by the HIFU beam path.
33. Any other reason for which the individual patient is not appropriate or suitable for participation.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Change in menstrual bleeding as measured by the Menstrual Pictogram (MP) score | At 12 months after treatment
  The Menstrual Pictogram (MP) is a validated pictorial instrument for measuring menstrual bleeding using modern superabsorbent sanitary products [6,7]. The MP score will be measured at 12 months after treatment and compared to the patient's baseline score to assess whether an improvement occurred. Success is defined for an individual patient as a ≥ 50% reduction in MP score from baseline or a final MP score ≤ 80 mL.
Rate of reintervention | At 12 months after treatment
  For the purposes of this study, reintervention refers to a procedure for the treatment of abnormal uterine bleeding related to fibroids other than a HIFU treatment using the Mirabilis System. A procedure is defined to include uterine artery embolization, endometrial ablation, radiofrequency ablation, cryotherapy, myomectomy, and hysterectomy. An additional treatment with the Mirabilis System as allowed by the protocol is not considered a reintervention. The rate of reintervention is defined as the percentage of patients who complete treatment with the Mirabilis System and subsequently undergo a different procedure for the treatment of abnormal uterine bleeding related to fibroids within 12 months after treatment. Success is defined for an individual patient as an absence of reintervention within this period.
Adverse event reports | Within 12 months after treatment
  The primary safety analysis will be performed on all patients receiving any HIFU treatment and will consist of a standardized assessment of all adverse events reported from the time that the patient's treatment starts until 12 months after treatment. The totality of safety information obtained from adverse event reports over this timeframe will be used to characterize the primary safety profile of the Mirabilis System via descriptive summaries.

SECONDARY OUTCOMES:
Change in Uterine Fibroid Symptom - Quality of Life (UFS-QOL) survey score | At 12 months after treatment
  The Uterine Fibroid Symptom - Quality of Life (UFS-QOL) survey is a validated and fibroid-specific assessment tool for measuring fibroid-related symptoms and their impact on the patient's quality of life [8]. The UFS-QOL survey score will be measured at 12 months after treatment and compared to the patient's baseline score to assess whether an improvement occurred. Because this is a secondary endpoint, the change in UFS-QOL survey score will be reported for informational purposes only, and there is no threshold for defining success in an individual patient.
Percentage of patients achieving pre-specified reductions in Menstrual Pictogram (MP) score | At 12 months after treatment
  The percentage of all patients completing treatment with the Mirabilis System who achieve pre-specified reductions in Menstrual Pictogram (MP) score at 12 months after treatment will be determined. These pre-specified reductions are: (1) percentage of patients achieving ≥ 22% reduction in MP score, (2) percentage of patients achieving ≥ 30% reduction in MP score, and (3) percentage of patients achieving ≥ 40% reduction in MP score. Because this is a secondary endpoint, these percentages of patients will be reported for informational purposes only, and there is no threshold for defining success for these percentages.
Change in treated fibroid volume as assessed by gadolinium-enhanced MRI | At 6 months after treatment
  The volume of each treated fibroid will be measured via gadolinium-enhanced MRI at 6 months after treatment and compared to its baseline volume also measured via gadolinium-enhanced MRI to assess whether fibroid shrinkage occurred. Because this is a secondary endpoint, the change in treated fibroid volume will be reported for informational purposes only, and there is no threshold for defining success in an individual patient.
Presence of newly-formed non-perfused volumes (NPV) in the targeted tissue | Within 72 hours after treatment
  The non-perfused volume (NPV) is the volume of tissue that no longer has blood flow as a result of treatment and is used as a marker of acute treatment effectiveness. The presence or absence of a newly-formed NPV (i.e., one that was not present prior to treatment) will be assessed via gadolinium-enhanced MRI within 72 hours after treatment. Because this is a secondary endpoint, the presence or absence of newly-formed NPVs will be reported for informational purposes only, and there is no NPV size threshold for defining success in an individual patient.
Adverse event reports | Within 24 months after treatment and within 36 months after treatment
  The secondary safety analysis will be performed analogously to the primary safety analysis on all adverse events reported within 24 months and within 36 months after treatment. The totality of safety information obtained from adverse event reports over these timeframes will be used to characterize the longer-term safety profile of the Mirabilis System via descriptive summaries.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lau, M.D., Study Director — Mirabilis Medica, Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parsons JE, Lau MPH, Martin PJ, Islas Lagos JJ, Aguilar Aguirre JM, Garza Leal JG. Pilot Study of the Mirabilis System Prototype for Rapid Noninvasive Uterine Myoma Treatment Using an Ultrasound-Guided Volumetric Shell Ablation Technique. J Minim Invasive Gynecol. 2017 May-Jun;24(4):579-591. doi: 10.1016/j.jmig.2017.01.010. Epub 2017 Jan 18. PMID 28109895
- [Background] Garza Leal JG, Hernandez Leon I, Castillo Saenz L, Aguilar Aguirre JM, Islas Lagos JJ, Parsons JE, Darlington GP, and Lau MPH. In-Office Rapid Volumetric Ablation of Uterine Fibroids under Ultrasound Imaging Guidance: Preclinical and Early Clinical Experience with the Mirabilis Transabdominal HIFU Treatment System. Proceedings of the 14th International Symposium on Therapeutic Ultrasound. AIP Conference Proceedings 1821: 020001 (2017).
- [Background] Garza Leal JG, Hernandez Leon I, Castillo Saenz L, Aguilar Aguirre JM, Islas Lagos JJ, Parsons JE, Martin PM, and Lau MPH. Refinement of the Shell Ablation Technique for Rapid In-Office Treatment of Uterine Fibroids under Ultrasound Imaging Guidance using the Mirabilis Transabdominal HIFU System. 15th International Symposium on Therapeutic Ultrasound Program and Abstracts: 156 (2015).
- [Background] Lau M, Aguilar Aguirre JM, Islas Lagos JJ, and Garza Leal JG. Office Based High-Speed Ultrasound Image Guided HIFU (High Intensity Focused Ultrasound) Ablation of Uterine Fibroids. Gynecol. Surg. 11 (Suppl. 1): 149-150 (2014).
- [Background] Garza Leal JG, Hernandez Leon I, Castillo Saenz L, Aguilar Aguirre JM, Islas Lagos JJ, Parsons JE, Darlington GP, and Lau MPH. In-Office Rapid Volumetric Ablation of Uterine Fibroids under Ultrasound Imaging Guidance: Preclinical and Early Clinical Experience with the Mirabilis Transabdominal HIFU Treatment System. 14th International Symposium on Therapeutic Ultrasound Program and Abstracts: 43 (2014).
- [Background] Magnay JL, Nevatte TM, O'Brien S, Gerlinger C, Seitz C. Validation of a new menstrual pictogram (superabsorbent polymer-c version) for use with ultraslim towels that contain superabsorbent polymers. Fertil Steril. 2014 Feb;101(2):515-22. doi: 10.1016/j.fertnstert.2013.10.051. Epub 2013 Dec 12. PMID 24331833
- [Background] Magnay JL, Nevatte TM, Seitz C, O'Brien S. A new menstrual pictogram for use with feminine products that contain superabsorbent polymers. Fertil Steril. 2013 Dec;100(6):1715-21.e1-4. doi: 10.1016/j.fertnstert.2013.08.028. Epub 2013 Sep 11. PMID 24034941
- [Background] Spies JB, Coyne K, Guaou Guaou N, Boyle D, Skyrnarz-Murphy K, Gonzalves SM. The UFS-QOL, a new disease-specific symptom and health-related quality of life questionnaire for leiomyomata. Obstet Gynecol. 2002 Feb;99(2):290-300. doi: 10.1016/s0029-7844(01)01702-1. PMID 11814511